CLINICAL TRIAL: NCT06871306
Title: Effects of Left and Bilateral Transcutaneous Auricular Vagus Nerve Stimulation on Pain, Mood, and Autonomic Function in Female Fibromyalgia Patients: A Randomized Controlled Trial
Brief Title: Effects of Left and Bilateral Transcutaneous Auricular Vagus Nerve Stimulation on Pain, Mood, and Autonomic Function in Female Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Burcu AKKURT, PHD, Fenerbahce University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 12.08.2021/31
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left taVNS (Active Comparator): Left taVNS group received taVNS stimulation through the left ear for 11 sessions.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Bilateral taVNS (Active Comparator): Bilateral taVNS group received taVNS stimulation through the bilateral ears for 11 sessions.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — taVNS was performed using the Vagustim device (Vagustim Health Technologies, Teknokent, Istanbul, Türkiye) at the tragus and concha regions for 30 minutes, with a frequency of 25 Hz and a pulse width of 300 µs in both groups. The difference in stimulation between the groups depends only on to which ear it was applied. Electrical stimulation was increased in 0.1 mA steps until the detection threshold was reached.

SUMMARY:
This study aimed to examine the effects of transcutaneous auricular vagus nerve stimulation (taVNS) on pain, depression, anxiety, functionality, and autonomic function in fibromyalgia syndrome (FMS).

primary hypothesis: TAVSS application is not an effective treatment for depression, physical limitation, functional disability, anxiety, pain and autonomic nerve system in female FMS patients.

secondary hypothesis: TAVSS application is an effective treatment for depression, physical limitation, functional disability, anxiety, pain and autonomic nerve system in female FMS patients.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteer participants
* Aged 18-45 with regular menstrual cycles
* Diagnosed with FMS (Widespread Pain Index≥ 17
* Symptom Severity Scale≥ 21) according to the 2013 ACR diagnostic criteria by a specialist physician.

Exclusion Criteria:

* Neurological deficits,
* Diabetes
* Neuropathic disorders
* Chronic inflammation
* Immune deficiencies
* Cardiac diseases
* Pregnancy
* Being in the perimenopausal or postmenopausal stages,
* Menstrual cycles of less than 28 days,
* Started new medication within the last 3 months,
* Modifications to their existing treatment apart from taVNS.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female participants are eligible for this study, as fibromyalgia syndrome is more prevalent in the female population.
Enrollment: 40 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | From enrollment to the 28th day of control
  Fibromyalgia Impact Questionnaire is a scale consisting of 10 questions, displaying physical function, absence from work, feeling well, fatigue, difficulty at work, pain, stillness, morning fatigue, anxiety, and depression. Apart from feeling well, low scores indicate recovery or being slightly affected by the disease. The maximum score of each subheading is 10 and the total score is 100. FIQ score was evaluated as being slightly affected under 50 points, moderately affected between 50-69, and heavily affected at 70 and more.
Visual Analog Scale | From enrollment to the 28th day of control
  Pain severity was assessed with the Visual Analog Scale (VAS), which is scored between 0 and 10, and is used to evaluate pain. 0 denotes no pain and 10 denotes unbearably severe pain. Participants were asked to mark the pain they felt on a 10 cm straight line and the value found was recorded in cm.
PNS Index Activity | From enrollment to the 28th day of control
  The PNS Index was used to measure ANS activity, indicating the evaluation of a person's parasympathetic nervous system activity compared to normal resting values. (https://www.kubios.com/publications/) The PNS index serves as a quantitative indicator of ANS function by reflecting the activity levels of its branches. This measures play a crucial role in heart rate variability (HRV) analysis, offering valuable insights into an individual's stress levels and recovery capacity. For PNS activity reduces heart rate and enhances HRV. HRV changes in pathological conditions (ischemic heart disease etc.), and decreased variability is a predictor of worse outcomes. Cyclical fluctuations in heart rate reveal changes in the ANS. The e-motion Faros device has been classified as a Class II medical device by Health Canada. After recording the R-R intervals of heart rate by e-motion Faros, the data were transferred to Kubios software for interpretation of HRV.
SNS Index Activity | From enrollment to the 28th day of control
  The SNS Index was used to measure ANS activity, indicating the evaluation of a person's sympathetic nervous system activity compared to normal resting values. (https://www.kubios.com/publications/) The SNS index serves as a quantitative indicator of ANS function by reflecting the activity levels of its branches. This measures play a crucial role in heart rate variability (HRV) analysis, offering valuable insights into an individual's stress levels and recovery capacity. A heightened SNS index is often associated with increased sympathetic activity, commonly linked HRV changes in pathological conditions (ischemic heart disease etc.), and decreased variability is a predictor of worse outcomes. Cyclical fluctuations in heart rate reveal changes in the ANS. The e-motion Faros device has been classified as a Class II medical device by Health Canada. After recording the R-R intervals of heart rate by e-motion Faros, the data were transferred to Kubios software for interpretation of HRV.
Assessment of Autonomic Nervous System Activity (SNS and PNS Index) | From enrollment to the 28th day of control
  Autonomic nervous system (ANS) activity, including both sympathetic (SNS) and parasympathetic (PNS) indices, is assessed using the eMotion Faros device. The device continuously records electrocardiographic (ECG) signals via a single-lead chest electrode setup. It is classified as a Class II medical device by Health Canada.
  The collected ECG data are analyzed using proprietary Kubios HRV Premium software, which computes time-domain, frequency-domain, and nonlinear heart rate variability (HRV) parameters. SNS and PNS indices are derived using Kubios' built-in algorithms that combine spectral analysis (e.g., LF/HF ratio), stress index, and other HRV-derived metrics to estimate autonomic balance.
  Higher SNS index values indicate increased sympathetic activity, while higher PNS index values reflect enhanced parasympathetic tone.

SECONDARY OUTCOMES:
Beck Depression Index | From enrollment to the 28th day of control
  The Beck Depression Index (BDI) is an evaluation questionnaire that assesses, behavioral signs of depression in adolescents and adults. The total score ranges from 0 to 63. It is interpreted as Minimal =0-9, Mild=10-16, Moderate=17-29 and Severe=30-63.
Beck Anxiety Inventory | From enrollment to the 28th day of control
  The Beck Anxiety Inventory (BAI) is suggested as a tool for evaluating clinical anxiety and distinguishing between anxious and non-anxious diagnostic groups. It is a 21-item Likert-type scale, scored from 0 to 3. The total score ranges from 0 to 63, with the following classifications: mild <21, moderate: 22-35, and severe>36

CONTACTS AND LOCATIONS:
Locations (1):
- Sancak Tıp Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.

REFERENCES:
- [Derived] Akkurt MF, Ozden AV, Akkurt HE, Akkurt B, Bildik C. Effects of left and bilateral transcutaneous auricular vagus nerve stimulation on pain, mood, and autonomic nervous system in female patients with fibromyalgia: a randomized controlled trial. Physiother Theory Pract. 2025 Dec 2:1-11. doi: 10.1080/09593985.2025.2594572. Online ahead of print. PMID 41332177